Efficacy and safety of ethanol inhalation on COVID-19 treatment (a clinical trial study)

IRCT registration number: IRCT20210725051981N1

**December 1, 2021** 

## **Statistical Analysis**

Based on the "treatment-on" or "protocol per" strategy, analysis was limited to participants who, according to the study protocol and inclusion criteria, received full interventions and informed the outcomes. Quantitative and qualitative variables were reported in the form of descriptive statistics including mean standard deviation and number (%), respectively. Quantitative variables with normal and abnormal distributions were compared between groups using independent t-test and Mann-Whitney test, respectively. In addition, qualitative variables were compared between the two groups using Chi-square test.

Comparisons between SPO2 values and clinical symptom scores on days 1, 3, 7 and 14 were performed using a mixed model. Mean changes of baseline values were measured by repeated measures analysis. The sphericity hypothesis was rejected with the help of Mauchly's Statistics and Geisser-Greenhouse correction was used for this purpose.

The proportion of patients who needed additional medical care after 14 days was tested in two groups using  $\chi 2$  test.

All statistical analyzes were performed using SPSS software version 22 (SPSS Inc., Chicago, IL, USA) and P < 0.05 was considered significant.